CLINICAL TRIAL: NCT04457622
Title: Language and Brain Rhythms
Acronym: LaBRhythms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL20_0333; 2020-A01231-38 (Other: ID-RCB)
Record Dates: First submitted 2020-06-12; First posted 2020-07-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
Keywords: Auditory Perception; Speech; Neuroimaging
MeSH Terms: conditions — Speech

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main study group (Experimental): All participants signed up for experiment 1, 2, 3 or 4 complete the same protocol (1 study arm) with an intent for intra-subject correlational analyses
  Interventions: Other: Auditory perception tasks in healthy participants

INTERVENTIONS:
Other: Auditory perception tasks in healthy participants — The participants complete auditory perception tasks while EEG, and MEG record brain signals (primary outcome measure). The tasks acquire behavioral responses with button presses (secondary outcome measure).
  All analyses are intra-subject (no analyses are between-subject).

SUMMARY:
For humans and other animals, predicting the timing of sensory events is essential for their daily behavior. Importantly, natural sensory stimulation (such as movements, music, or speech) can present temporal regularities allowing for temporal prediction of incoming sensory information. For instance, individuals can easily predict in time the next step of a walker, or the next beat of a song based on the rhythm. The phenomenon of temporal prediction has for now only been investigated experimentally in deterministic scenarios, i.e. when the duration between two sensory events is fixed, or when stimuli present a regular beat. The objective of this project is to understand how we process more natural, hence more complex forms of temporal regularities, and how individuals make inferences on the timing of sensory events based on past temporal statistics of sensory information. This is particularly important for speech processing, considering that speech is an acoustic signal that is known to possess some form of temporal regularity, and yet is not purely rhythmic nor does have a deterministic temporal structure. Temporal regularities are specific to each spoken language, and both native and non-native language listeners are known to use temporal acoustic cues during speech listening. This affects speech comprehension and has a strong impact during language learning. Hence, understanding the processing of temporal regularities in speech can help improve language abilities in first and second language learners.

The project is composed of four experiments. The first behavioral experiment will investigate how auditory perception is affected by the temporal statistics of past sensory information using artificial stimuli. The second axis will investigate the neural mechanisms underlying auditory timing processing with electroencephalography (EEG). The last Magnetoencephalography (MEG, experiment 3) and EG (rxperiement 4) experiment will test the role of temporal statistics in an ecological setting, namely speech listening. The project will thus provide strong theoretical advances as it will give new insights on brain mechanisms for the processing of complex temporal information in audition and speech, and their role in language comprehension. It will also provide methodological advances. Specifically, the project will contribute to the development and validation of cutting-edge methods in MEG. Namely, it will aim at creating new tools to investigate the neural correlates of auditory and speech processing with an unprecedented temporal and spatial resolution.

ELIGIBILITY:
Inclusion Criteria:

For all experiments:

* 18- 40 years old
* Registration with the French healthcare system
* Informed consent
* Normal hearing

Additionally, for experiments 2,3 and 4 :

- Right handed

Additionally, for experiment 3 and 4:

- French as native language

Exclusion Criteria:

For All Experiments:

* Neurological or psychiatric illnesses or a history of such problems that could impact quality/variability of data or cooperation and retention of the subject in the study
* Regular use of medications that impact the central nervous system
* Regular use of medications, such as opioids and antidepressants, including SSRIs and tricyclic antidepressants
* Severe hearing loss
* A history of stroke or recent trauma to the head
* Persons unable to adhere to abstinence from the use of drugs or alcohol the day or evening before experimental sessions
* Women who are pregnant, breastfeeding, or have given birth in the last 6 months

Additionally, for experiment 2,3 and 4 :

* A pacemaker, insulin or other pump, neurostimulator, cochlear implants or other hearing aid, metal stents, prosthesis, or implants, intracerebral clips, implantable defibrillator, cerebral shunt or ventricular catheter, other foreign metal objects in the upper part of the body
* any dental apparatus containing metal including or root canals
* any foreign metallic object anywhere in the body
* bolts, screws
* orthopedic devices or implants

Additionally, for experiment 3 and 4:

* claustrophobia
* glasses (given the participant cannot use contact lenses)
* a head size incompatible with the use of a personalized 3D headcast or a magnetoencephalography
* Persons having had any surgery prior to the study which puts them at risk for metal objects left in the body

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 356 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2026-10-18 (Estimated); Study Completion 2026-10-18 (Estimated)

PRIMARY OUTCOMES:
Stimulus-Brain (EEG) Coherence in the delta-theta range (1 Hz - 8 Hz) | at max 90 days
Amplitude of EEG evoked responses to the target stimuli | at max 90 days
Stimulus-Brain (MEG) Coherence in the delta-theta range (1 Hz - 8 Hz) | at max 90 days
Amplitude of MEG evoked responses to the target stimuli | at max 90 days

SECONDARY OUTCOMES:
Percentage of correct responses | at max 90 days
  The secondary outcome measures will be recorded in all experiments
Response Times | at max 90 days
  The secondary outcome measures will be recorded in all experiments

CONTACTS AND LOCATIONS:
Overall Officials: Anne KOSEM, PhD, Principal Investigator — Centre de recherche de Neurosciences de Lyon (CRNL)
Locations (1):
- Centre de Recherche en Neuroscience de Lyon, Bron, France